CLINICAL TRIAL: NCT01000662
Title: Phase III Study Comparing Whole Breast Radiotherapy With a Daily Tumor Red Boost
Brief Title: Study Comparing Whole Breast Radiotherapy With a Daily Versus a Weekly Tumor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09-0030
Record Dates: First submitted 2009-10-09; First posted 2009-10-23 (Estimated); Results first posted 2015-05-29 (Estimated); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
Keywords: whole breast radiotherapy; tumor bed boost
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ARM 1 daily boost (Active Comparator): Radiation Therapy
  Interventions: Radiation: Daily Radiation Therapy
- ARM 2 weekly boost (Active Comparator): Radiation Therapy
  Interventions: Radiation: Weekly Radiation Therapy

INTERVENTIONS:
Radiation: Daily Radiation Therapy — 15 daily radiation fractions of 2.7 Gy, Monday to Friday for 3 weeks, to the whole breast with a daily concomitant boost of 0.5 Gy to the tumor bed, for a total daily dose of 3.2 Gy to the tumor bed (2.7Gy+0.5 Gy). The overall dose will be 40.5 Gy to the breast and 48.0 Gy to the tumor bed.
  Arms: ARM 1 daily boost
Radiation: Weekly Radiation Therapy — 15 weekly radiation fractions of 2.7 Gy Monday to friday for three weeks to the entire breast with a Friday boost of 2.0 Gy to the tumor bed, for a total dose to the tumor bed on each friday of 4.7 Gy (2.7 Gy+ 2.0 Gy). The overall dose will be 40.5 Gy to the breast and 46.5 gy to the tumor bed.
  Arms: ARM 2 weekly boost

SUMMARY:
All patients (with Stages 0-II breast cancer) will receive an accelerated three week regimen of prone whole breast radiotherapy. The study intends to test the hypothesis that a weekly boost to the tumor bed, delivered on Friday, before the weekend break, is as well tolerated as the daily boost during accelerated prone radiotherapy.

DETAILED DESCRIPTION:
Arm 1 is a concomitant boost protocol over three weeks which has previously been evaluated in over 500 patients (NYU 03-30 and NYU 05-181) and has shown excellent tolerance, and results. Arm 2 evaluates a Weekend Boost Dose (WBD) regimen which may have a radiobiological advantage by counteracting tumor repopulation which can occur over the weekend break. At the time of registration in the study, patients will be randomized to either treatment arm and stratified according to pre or post-menopausal status and on previous chemotherapy received or not.

ELIGIBILITY:
Inclusion Criteria:

* Pre or post-menopausal women with stage 0,I, and II breast cancer
* Biopsy-proven invasive breast cancer, excised with negative margins of at least 1 mm
* Status post segmental mastectomy, after sentinel node biopsy and/or axillary node dissection (DCIS and Tumors <5mm do not require nodal assessment)
* At least 2 weeks from last chemotherapy
* Patient needs to be able to understand and demonstrate willingness to sign a written informed consent document

Exclusion Criteria:

* Previous radiation therapy to the ipsilateral breast
* More than 3 involved nodes identified at axillary staging, requiring adjuvant axillary radiation
* Active connective tissue disorders, such as lupus or scleroderma
* Prior or concurrent malignancy other than basal or squamous cell skin cancer or carcinoma in-situ of the cervix, unless disease-free >3 years
* Pregnant or lactating women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2009-03; Primary Completion 2012-07 (Actual); Study Completion 2017-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Perez, MD, Principal Investigator — NYU School of Medicine
Locations (3):
- United States (3):
  - Bellevue Hospital Center, New York, New York
  - NYU Clinical Cancer Center, New York, New York
  - Tisch Hospital, New York, New York

REFERENCES:
- [Result] Cooper BT, Formenti-Ujlaki GF, Li X, Shin SM, Fenton-Kerimian M, Guth A, Roses DF, Hitchen CJ, Rosenstein BS, Dewyngaert JK, Goldberg JD, Formenti SC. Prospective Randomized Trial of Prone Accelerated Intensity Modulated Breast Radiation Therapy With a Daily Versus Weekly Boost to the Tumor Bed. Int J Radiat Oncol Biol Phys. 2016 Jun 1;95(2):571-8. doi: 10.1016/j.ijrobp.2015.12.373. Epub 2015 Dec 29. PMID 27131077
- [Result] Garsa AA, Ferraro DJ, DeWees TA, Deshields TL, Margenthaler JA, Cyr AE, Naughton M, Aft R, Gillanders WE, Eberlein T, Matesa MA, Ochoa LL, Zoberi I. A prospective longitudinal clinical trial evaluating quality of life after breast-conserving surgery and high-dose-rate interstitial brachytherapy for early-stage breast cancer. Int J Radiat Oncol Biol Phys. 2013 Dec 1;87(5):1043-50. doi: 10.1016/j.ijrobp.2013.09.009. Epub 2013 Oct 22. PMID 24161428
- [Derived] Finkel MA, Cooper BT, Li X, Fenton-Kerimian M, Goldberg JD, Formenti SC. Quality of Life in Women Undergoing Breast Irradiation in a Randomized, Controlled Clinical Trial Evaluating Different Tumor Bed Boost Fractionations. Int J Radiat Oncol Biol Phys. 2016 Jun 1;95(2):579-89. doi: 10.1016/j.ijrobp.2016.02.004. Epub 2016 Feb 6. PMID 27045811

RESULTS

PARTICIPANT FLOW:
Groups:
- ARM 1 Daily Boost: Radiation Therapy
  15 daily radiation fractions of 2.7 Gy, Monday to Friday for 3 weeks, to the whole breast with a daily concomitant boost of 0.5 Gy to the tumor bed, for a total daily dose of 3.2 Gy to the tumor bed (2.7Gy+0.5 Gy). The overall dose will be 40.5 Gy to the breast and 48.0 Gy to the tumor bed.
- ARM 2 Weekly Boost: Radiation Therapy
  15 weekly radiation fractions of 2.7 Gy Monday to friday for three weeks to the entire breast with a Friday boost of 2.0 Gy to the tumor bed, for a total dose to the tumor bed on each friday of 4.7 Gy (2.7 Gy+ 2.0 Gy). The overall dose will be 40.5 Gy to the breast and 46.5 gy to the tumor bed.
Period: Overall Study
Arm/Group | ARM 1 Daily Boost | ARM 2 Weekly Boost
Started | 206 | 206
Completed | 202 | 198
Not Completed | 4 | 8

BASELINE CHARACTERISTICS:
Groups:
- ARM 1 Daily Boost; ARM 2 Weekly Boost: Radiation Therapy
  Radiation Therapy: Arm 1= 15 daily radiation fractions of 2.7 Gy, Monday to Friday for 3 weeks, to the whole breast with a daily concomitant boost of 0.5 Gy to the tumor bed, for a total daily dose of 3.2 Gy to the tumor bed (2.7Gy+0.5 Gy). The overall dose will be 40.5 Gy to the breast and 48.0 Gy to the tumor bed.
  Arm 2= 15 daily radiation fractions of 2.7 Gy Monday to friday for three weeks to the entire breast with a Friday boost of 2.0 Gy to the tumor bed, for a total dose to the tumor bed on each friday of 4.7 Gy (2.7 Gy+ 2.0 Gy). The overall dose will be 40.5 Gy to the breast and 46.5 gy to the tumor bed.
- Total: Total of all reporting groups
Arm/Group | ARM 1 Daily Boost | ARM 2 Weekly Boost | Total
Number analyzed (Participants) | 206 | 206 | 412
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 155 | 168 | 323
  >=65 years | 51 | 38 | 89
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 206 | 206 | 412
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 19 | 17 | 36
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 21 | 26 | 47
  White | 158 | 150 | 308
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 13 | 19
Region of Enrollment [Number; unit: participants]
  United States | 206 | 206 | 412

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Radiation Toxicities Recorded According to Radiation Therapy Oncology Group (RTOG)
Description: Number of patients with a grade 2 or greater toxicity after 3 weeks of whole breast IMRT with a once/week boost compared to those patients treated with a daily boost: 0 - no symptoms, 5 - death directly related to radiation effects
Time Frame: Day 60
Population: Patients receiving either daily or weekly boost to radiation therapy
Measure: Number; unit: participants
Arm/Group | ARM 1 Daily Boost | ARM 2 Weekly Boost
Number analyzed (Participants) | 202 | 198
participants | 22 | 16

2. Secondary Outcome: Average Score on Breast Cancer Treatment Outcomes Scale (BCTOS) at Baseline
Description: BCTOS is a validated questionnaire designed to measure breast esthetic and function after breast-conservations treatment. Patients rate the difference between their untreated and treated breast in 3 categories.
  There are 4 score levels: 1 = "No difference"; 2 = "Slight"; 3 = "Moderate"; 4 = "Large difference". The total range is 3-12; the lower the score the lower the difference between the untreated and treated breast.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARM 1 Daily Boost | ARM 2 Weekly Boost
Number analyzed (Participants) | 202 | 198
score on a scale
  Functional Status | 6.89 (2.72) | 7.03 (2.74)
  Cosmetic Status | 9.71 (3.2) | 9.9 (3.32)
  Breast Specific Pain | 3.69 (1.28) | 3.87 (1.47)

3. Secondary Outcome: Score on "SF-36 v2 Vitality" Scale
Description: SF-36 is an extensively used questionnaire designed to compare health status across various populations and is commonly used in cancer trials Our survey includes the portion of the SF-36 focused on the assessment of patient fatigue, or "vitality," at various stages of treatment Example question: How much of the time during the past 4 weeks did you feel full of life? (Answer on scale 1 to 5). 1 = "All of the time"; 2 = "Most of the time"; 3 = "Some of the time"; 4 = "A little of the time"; 5 = "None of the time".
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARM 1 Daily Boost | ARM 2 Weekly Boost
Number analyzed (Participants) | 202 | 198
score on a scale
  Good Feeling | 2.56 (0.91) | 2.65 (0.95)
  Bad Feeling | 3.3 (0.88) | 3.3 (0.97)

4. Secondary Outcome: Average Score on Brief Pain Inventory (BPI) Scale
Description: The BPI is a self-administered assessment tool used in pain management.
  The BPI scale defines pain as follows:
  1-4 = Mild Pain 5-6 = Moderate Pain 7-10 = Severe Pain
  The total range is 1-10; the higher the score, the higher the pain level.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARM 1 Daily Boost | ARM 2 Weekly Boost
Number analyzed (Participants) | 202 | 198
score on a scale | 1.46 (1.59) | 1.71 (1.65)

5. Secondary Outcome: Average Score on Radiation Therapy Oncology Group (RTOG) Breast Quality of Life Scale
Description: 4 levels: 1 = "Excellent"; 2 = "Good"; 3 = "Fair"; 4 = "Poor." The total range is 1-4; the higher the score, the lower the breast quality.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARM 1 Daily Boost | ARM 2 Weekly Boost
Number analyzed (Participants) | 202 | 198
score on a scale
  Satisfaction on Breast Looks | 1.97 (0.78) | 1.96 (0.84)
  Satisfaction about Treatment | 1.47 (0.78) | 1.41 (0.71)
  Convenience of Care | 2.53 (2.38) | 2.84 (2.41)

6. Secondary Outcome: Average Score on Breast Cancer Treatment Outcomes Scale (BCTOS) at the End of Treatment
Description: as for outcome 2
Time Frame: At the end of Treatment, an average of 3 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARM 1 Daily Boost | ARM 2 Weekly Boost
Number analyzed (Participants) | 202 | 198
score on a scale
  Functional Status | 7.08 (2.72) | 7.56 (3.24)
  Cosmetic Status | 10.29 (3.17) | 10.10 (3.11)
  Breast Specific Pain | 4.57 (1.34) | 4.51 (1.51)

7. Secondary Outcome: Average Score on Breast Cancer Treatment Outcomes Scale (BCTOS)
Description: as for outcome 2
Time Frame: 45-60 days after treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARM 1 Daily Boost | ARM 2 Weekly Boost
Number analyzed (Participants) | 202 | 198
score on a scale
  Functional Status | 6.93 (3.13) | 7.01 (2.79)
  Cosmetic Status | 10.17 (3.07) | 10.00 (2.84)
  Breast Specific Pain | 3.94 (1.34) | 3.80 (1.40)

8. Secondary Outcome: Score on "SF-36 v2 Vitality" Scale
Description: as for outcome 3
Time Frame: End of Treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARM 1 Daily Boost | ARM 2 Weekly Boost
Number analyzed (Participants) | 202 | 198
score on a scale
  Good Feeling | 2.55 (0.87) | 3.59 (0.92)
  Bad Feeling | 3.32 (0.86) | 3.25 (0.99)

9. Secondary Outcome: Score on "SF-36 v2 Vitality" Scale 45-60 Days After Treatment
Description: as for outcome 3
Time Frame: 45-60 days after treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARM 1 Daily Boost | ARM 2 Weekly Boost
Number analyzed (Participants) | 202 | 198
score on a scale
  Good Feeling | 2.46 (0.78) | 2.36 (0.91)
  Bad Feeling | 3.29 (0.92) | 3.45 (0.84)

10. Secondary Outcome: Average Score on Brief Pain Inventory (BPI)
Description: as for outcome 4
Time Frame: At the end of Treatment, an average of 3 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARM 1 Daily Boost | ARM 2 Weekly Boost
Number analyzed (Participants) | 202 | 198
score on a scale | 1.46 (1.59) | 1.66 (1.67)

11. Secondary Outcome: Average Score on Brief Pain Inventory (BPI)
Description: as for outcome 4
Time Frame: 45-60 days after treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARM 1 Daily Boost | ARM 2 Weekly Boost
Number analyzed (Participants) | 202 | 198
score on a scale | 1.23 (1.51) | 1.37 (1.52)

12. Secondary Outcome: Score on Radiation Therapy Oncology Group (RTOG) Breast Quality of Life Scale, at End of Treatment
Description: 4 levels: 1 = "Excellent"; 2 = "Good"; 3 = "Fair"; 4 = "Poor"
Time Frame: End of Treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARM 1 Daily Boost | ARM 2 Weekly Boost
Number analyzed (Participants) | 202 | 198
score on a scale
  Breast Looks now | 2.12 (0.74) | 1.95 (0.82)
  Satisfaction about Treatment | 1.35 (0.68) | 1.33 (0.65)

13. Secondary Outcome: Score on Radiation Therapy Oncology Group (RTOG) Breast Quality of Life Scale, 45-60 Days After Treatment
Description: 4 levels: 1 = "Excellent"; 2 = "Good"; 3 = "Fair"; 4 = "Poor."
Time Frame: 45-60 days after treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARM 1 Daily Boost | ARM 2 Weekly Boost
Number analyzed (Participants) | 202 | 198
score on a scale
  Breast Looks now | 2.02 (0.73) | 1.94 (0.76)
  Satisfaction about Treatment | 1.33 (0.72) | 1.32 (0.67)

ADVERSE EVENTS:
Time Frame: Day 1 of radiation therapy to Day 60
Arm/Group | ARM 1 Daily Boost | ARM 2 Weekly Boost
Serious Adverse Events (participants affected / at risk) | 0/202 | 0/198
Other Adverse Events (participants affected / at risk) | 89/202 | 72/198
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM 1 Daily Boost (N=202) | ARM 2 Weekly Boost (N=198)
Edema (Grade 1) (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Fibrosis (Grade 1) (Reproductive system and breast disorders) | 26 (28) | 17 (17)
Pain (Grade 1) (Reproductive system and breast disorders) | 10 (10) | 12 (12)
Pigmentation Change (Grade 1) (Skin and subcutaneous tissue disorders) | 15 (18) | 13 (13)
Retraction/Atrophy (Grade 1) (Skin and subcutaneous tissue disorders) | 23 (25) | 23 (23)
Telangiectasia (Grade 1) (Skin and subcutaneous tissue disorders) | 13 (13) | 4 (4)
Lymphedema (Grade 1) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No